CLINICAL TRIAL: NCT02451800
Title: Exercise: Improving Compliance and Long-term Weight Loss With Sanford Profile Program
Brief Title: Exercise: Improving Compliance and Long-term Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1411008
Record Dates: First submitted 2015-01-30; First posted 2015-05-22 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- in-class yoga (Experimental): The intervention is a in-class yoga course taught by yoga instructors for 3 times per week for 3 months. This class is based on "Peggy Cappy's Program: More Yoga for Every Body". Class is taught at Sanford Wellness Centers in Sioux Falls, South Dakota and Fargo, North Dakota. Each class in 1 hour in length.
  Interventions: Other: in-class yoga
- yoga by DVD (Active Comparator): For the intervention participants are asked to do yoga at home following the "Peggy Cappy's Program: More Yoga for Every Body" DVD. They are asked to complete these exercises 3 times per week for 3 months. The DVD is 1 hour in length.
  Interventions: Other: yoga by DVD
- stretching by DVD (Active Comparator): For the intervention participants are asked to do stretching exercises at home following "Bob Anderson's DVD-Stretching: the DVD". They are asked to complete these exercises 3 times per week for 3 months. The DVD is 1 hour in length.
  Interventions: Other: stretching by DVD

INTERVENTIONS:
Other: in-class yoga — In-person yoga classes that meet for 3x/week for 3 months. Each class is 1 hour.
  Arms: in-class yoga
Other: yoga by DVD — Individuals are asked to follow a 1-hour DVD on yoga 3x/week for 3 months.
  Arms: yoga by DVD
Other: stretching by DVD — Individuals are asked to follow a 1-hour DVD on stretching exercises 3x/week for 3 months.
  Arms: stretching by DVD

SUMMARY:
The overall aim of the proposed study is to determine the effectiveness of a 3-month yoga program on increasing compliance and improving weight loss while participating in the Sanford Profile program. Participants are randomized to one of three groups: in-class yoga, yoga by digital video disk (DVD), stretching by DVD. Changes in weight loss and stress levels are monitored.

DETAILED DESCRIPTION:
The overall aim of the proposed study is to determine the effectiveness of a 3-month yoga program on increasing compliance and improving weight loss while participating in the Sanford Profile program. The 6-month study includes a 3-month randomized, controlled trial using in-person yoga, a yoga DVD, and a stretching DVD (control group) followed by a 3-month post-intervention follow-up. The study will be conducted to test the hypotheses that both in-person yoga classes and DVD yoga participation will result in 1) greater compliance with the Profile program, 2) greater weight loss during the yoga intervention, and 3) greater weight loss 3 months following completion of the intervention compared to the stretching intervention. Compliance will be investigated using percent of days that dietary intake was entered online and percent of days that online records indicate that the program was followed. Changes in weight will be measured using data transmitted from electronic scales that are provided as part of the Profile program. In order to assess weight change after participation in the intervention we will ask participants to continue weighing themselves daily for 3 months following completion of the intervention regardless of whether they completed the Profile program or not. Participants will complete online questionnaires on behavioral and appetite perceptions related to eating, food intake, stress levels, compliance with diet recommendations given to them by Sanford Profile, and perceived benefits of their intervention. We will use these measures to determine the effect of yoga participation on eating behaviors and stress levels.

ELIGIBILITY:
Inclusion Criteria:

* Must be participants in the Sanford Profile Program (weight loss program)

Exclusion Criteria:

* Must have physician approval if answers yes to Physical Activity Readiness Questionnaire (PARQ) questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3 months
  All participants are enrolled in a weight loss program. This outcome will tell us whether yoga increases weight loss during the intervention.

SECONDARY OUTCOMES:
Weight loss | 6 months
  This outcome will tell us whether yoga participation results in long-term weight loss 3 months after the intervention stops.
Stress levels | 3 months
  Stress levels are measured using the Perceived Stress Scale (PSS). This outcome will tell us whether yoga participation reduces stress levels during intervention.
Stress levels | 6 months
  Stress levels are measured using the Perceived Stress Scale (PSS). This outcome will tell us whether yoga participation has a long-term (3 mo) effect on reducing stress after intervention stops.

CONTACTS AND LOCATIONS:
Overall Officials: Bonny L Specker, PhD, Study Director — South Dakota State University
Locations (1):
- South Dakota State University, Brookings, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No